CLINICAL TRIAL: NCT07272096
Title: Randomised Controlled Trial for a Novel ACT-based Videogame 'ACTing Minds' to Support Mental Health
Brief Title: ACTing Minds: An ACT-based Videogame for Mental Health
Acronym: ACTingMindsRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Darren Edwards, Associate Professor, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-PSY-ACTM-RCT-01
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Depression; Anxiety; Stress (Psychology); Psychological Flexibility; Quality of Life; Social Connectedness; Wellbeing
Keywords: Acceptance and Commitment Therapy; ACT; Psychological flexibility; Digital mental health; Serious game; Videogame intervention; Single-session intervention; Randomised controlled trial; CompACT; DASS-21; Flourishing Scale; Social Connectedness Scale; EQ-5D; Heart rate variability; HRV; ECG
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm, 1:1 randomised, single-session, laboratory-based trial.
Who Masked: Participant
Masking Description: Participants masked to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTing Minds (ACT videogame) (Experimental): Single ~60-minute session on a study-supplied smartphone in the lab; assessments at baseline, post-session, and short-term follow-up (10-13 days post-intervention).
  Interventions: Behavioral: ACTing Minds (ACT videogame)
- Neutral commercial puzzle game (Monument Valley) (Active Comparator): Engagement- and time-matched ~60-minute smartphone session in the lab; assessments at baseline, post-session, and short-term follow-up (10-13 days post-intervention).
  Interventions: Behavioral: Monument Valley (mobile; neutral control)

INTERVENTIONS:
Behavioral: ACTing Minds (ACT videogame) — Single-session (~60 min) ACT-based videogame integrating acceptance/openness, cognitive defusion, present-moment awareness, values and values-guided action via structured chapters. Delivered on a study-supplied Samsung Galaxy S9+ (Android) under standardised instructions; no therapist guidance during play.
  Arms: ACTing Minds (ACT videogame)
Behavioral: Monument Valley (mobile; neutral control) — Commercial mobile puzzle game used as an engagement- and time-matched control (~60 min) with no therapeutic content. Delivered on a study-supplied Samsung Galaxy S9+ (Android) in the lab. Title/version fixed for the trial; procedures and environment identical to the experimental arm. No data are collected within the app.
  Arms: Neutral commercial puzzle game (Monument Valley)

SUMMARY:
The goal of this clinical trial is to test whether a single-session Acceptance and Commitment Therapy (ACT) videogame (ACTing Minds) improves psychological flexibility and mental health in adults who report mild to moderate depression, anxiety or stress. The main questions are whether ACTing Minds increases psychological flexibility (CompACT Total) more than a time- and engagement-matched neutral commercial game at the end of the session and again at short-term follow-up (10-13 days), and whether it produces favourable changes in symptoms, wellbeing, social connectedness, health-related quality of life, and short seated heart-rate variability recordings. Researchers will compare ACTing Minds with the neutral game to determine whether the ACT-based experience leads to greater improvements. Participants attend one laboratory visit of about 60 minutes, complete brief questionnaires at baseline, immediately after the session and at short-term follow-up, and provide a short seated ECG at each timepoint for heart-rate variability analysis. The study uses a single-blind, two-arm, randomised, parallel-group design at Swansea University (UK).

DETAILED DESCRIPTION:
This trial evaluates a brief, scalable approach to supporting common mental health difficulties by embedding Acceptance and Commitment Therapy (ACT) processes in an engaging interactive experience. ACT targets psychological flexibility, the capacity to make values-guided choices while openly contacting difficult thoughts and feelings. ACTing Minds integrates core ACT processes (openness and acceptance, cognitive defusion, present-moment awareness, values clarification and values-guided action) within a structured, single-session videogame.

The objective is to determine whether ACTing Minds yields greater improvement in psychological flexibility and psychological distress than a neutral, engagement-matched game, and whether those process-level changes are accompanied by improvements in wellbeing and related functioning. The trial specifies two co-primary outcomes: psychological flexibility, assessed with the CompACT total score, and general psychological distress, assessed with the DASS-21 total score. For each co-primary outcome, the prespecified primary estimand is the between-group difference in change from baseline to short-term (10-13 days) follow-up. Secondary estimands examine change in CompACT and DASS-21 subscales, subjective wellbeing, social connectedness, health-related quality of life, and autonomic regulation indexed by heart-rate variability derived from short seated ECG recordings.

The study uses a two-arm, parallel-group, randomised design with 1:1 allocation at a single university laboratory site. Randomisation is computer-generated with concealed allocation and implemented after baseline assessment to prevent foreknowledge of assignment. Participants are masked to condition, and blinding integrity is assessed at follow-up by asking participants to guess their allocation. Both arms follow identical procedures and time on task; the comparator is a neutral commercial game selected to match the ACT intervention for duration and engagement while avoiding therapeutic content.

Assessments occur at baseline, immediately after the single session, and 10-13 days post-intervention. Questionnaires are administered electronically with built-in range and completeness checks to minimise entry errors. ECG is recorded seated for about five minutes per timepoint (Lead II). Heart-rate variability processing follows standard steps: signal inspection, identification and correction of artefacts, R-peak verification, derivation of time- and frequency-domain indices, and natural-log transformation of skewed metrics prior to modelling. Mean heart rate (beats per minute) is retained to contextualise autonomic indices.

The statistical analysis plan is specified as follows. Primary and secondary outcomes will be analysed using linear mixed-effects models with fixed effects of Condition, Timepoint and their interaction, and a random intercept for participant to accommodate within-person correlation and incomplete follow-up under maximum likelihood. Residual covariance structures (for example, autoregressive versus unstructured) will be compared using information criteria, retaining the better-fitting specification for each outcome family. The primary contrasts estimate group differences in change from baseline to short-term follow-up on the two co-primary outcomes, CompACT Total and DASS-21 Total; post-session contrasts and 95% confidence intervals will also be reported. Heart-rate variability variables will be analysed on the natural-log scale. Two-sided tests with an alpha of .05 will be used, with attention to confidence intervals and effect sizes. Analyses follow an intention-to-treat principle using all available data; planned sensitivity checks will include alternative covariance structures and, if warranted, supplementary multiple-imputation analyses for outcomes with materially higher missingness.

Data quality procedures include scripted data pipelines with version control, reproducible derivation of analysis datasets from raw sources, and automated checks for ranges, outliers and internal consistency across timepoints. The research team maintains a study data dictionary that defines each variable, coding and scoring rules, and any transformations applied. Access to identifiable data is role-based and restricted to authorised personnel; de-identified analysis files are stored on secure university systems. Adverse events are monitored during the laboratory session and at follow-up, and any serious events are managed according to institutional policy. Given the single-session, minimal-risk behavioural design, an independent data monitoring committee is not required.

The target sample size is approximately 300 participants, providing precise estimates of group differences and allowing robust sensitivity analyses. On completion of the trial and after primary publication, de-identified individual participant data, a data dictionary and analysis code will be shared on a public repository, subject to ethical and legal safeguards. Findings will be disseminated through peer-reviewed publications, conference presentations and lay summaries suitable for non-specialist audiences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to read and understand English
* Self-reported mild to moderate symptoms of depression, anxiety, or stress
* Provides written informed consent
* Willing and able to attend one ~60-minute laboratory session and complete online follow-up questionnaires 10-13 days later
* Agrees to ECG recording (seated ~5 minutes at each timepoint)
* Willing to play either study videogame on a study-supplied Samsung Galaxy S9+ (Android)

Exclusion Criteria:

* Current or past severe mental illness (e.g., psychotic disorder, bipolar disorder)
* Current psychotropic medication use (e.g., antidepressants, anxiolytics, antipsychotics, mood stabilisers, stimulants)
* Concurrent psychological therapy (any modality)
* Pregnancy
* Cardiovascular conditions or clinically significant arrhythmias that could affect ECG or HRV measurement or be exacerbated by study procedures
* Implanted cardiac devices (e.g., pacemaker or ICD)
* Any neurological condition, medical condition, or skin condition that would preclude safe ECG electrode placement or comfortable seated recording
* Insufficient English proficiency to provide informed consent or complete study measures
* Any other factor that, in the judgement of the investigators, would compromise safety, data quality, or protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2025-11-26 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Psychological flexibility (CompACT Total) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); short-term follow-up (10-13 days post-intervention).
  CompACT total score; higher scores indicate greater psychological flexibility. Primary estimand is the between-group difference in change from baseline to short-term follow-up (10-13 days post-intervention); post-session estimates will also be reported.
Mental-health symptoms (DASS-21 Total) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  DASS-21 total score; higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Depressive symptoms (DASS-21 Depression) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  DASS-21 Depression subscale; higher scores indicate greater depressive symptoms.
Anxiety symptoms (DASS-21 Anxiety) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  DASS-21 Anxiety subscale; higher scores indicate greater anxiety symptoms.
Stress symptoms (DASS-21 Stress) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  DASS-21 Stress subscale; higher scores indicate greater stress.
Wellbeing (Flourishing Scale) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Flourishing Scale total score; higher scores indicate greater psychological wellbeing.
Social connectedness (Social Connectedness Scale) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Social Connectedness Scale total score; higher scores indicate a stronger sense of connectedness/belonging.
Health-related quality of life (EQ-5D Index) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  EQ-5D index score derived from health state profiles; higher values indicate better health status.
Self-rated health (EQ-5D Visual Analogue Scale) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  EQ-5D VAS (0-100); higher values indicate better perceived health.
Heart-rate variability - lnRMSSD | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Natural-log root mean square of successive differences from 5-minute seated ECG; higher values reflect greater short-term HRV.
Heart-rate variability - lnSDNN | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Natural-log standard deviation of normal-to-normal intervals from 5-minute seated ECG.
Heart-rate variability - lnHF power | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Natural-log high-frequency power (conventional HF band) from 5-minute seated ECG.
Heart-rate variability - lnLF power | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Natural-log low-frequency power (conventional LF band) from 5-minute seated ECG.
Heart-rate variability - ln(LF/HF) ratio | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Natural-log LF/HF ratio from 5-minute seated ECG.
Mean heart rate (beats per minute) | Baseline (Day 0); Immediately post-intervention (≈60 minutes after Baseline); Short-term follow-up (10-13 days post-intervention).
  Mean heart rate recorded alongside ECG at each timepoint to contextualise HRV analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Darren J Edwards, PhD, Principal Investigator — Swansea University
Locations (1):
- Swansea University, School of Psychology (Singleton Park), Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data (IPD) underlying the published results, including all questionnaire outcomes (CompACT total/subscales, DASS-21 total/subscales, Flourishing, Social Connectedness, EQ-5D index and VAS), heart-rate variability summary indices (lnRMSSD, lnSDNN, lnHF, lnLF, lnLF/HF) and mean heart rate at T1-T3, allocation group, age band and gender. A data dictionary, statistical analysis plan and analysis code will be provided. Raw ECG waveforms and any free-text fields will not be shared. Data will be deposited on the Open Science Framework and released at article acceptance/publication; access will be open (no application) under an appropriate licence.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and documents will be made available at article acceptance/publication. If journal processes impose a brief embargo, release will occur within 3 months of acceptance. Materials will be retained indefinitely with versioning; any material updates (e.g., errata, code revisions) will be posted to the same repository. The registry will be updated with the dataset DOI/URL on release.
Access Criteria: Open access: no application required. De-identified IPD (questionnaire outcomes, HRV summary indices, mean heart rate, allocation group, age band, gender), data dictionary, SAP, protocol, consent template, and analysis code will be downloadable from a public repository.

REFERENCES:
- [Background] Edwards DJ, Kemp AH. A novel ACT-based video game to support mental health through embedded learning: a mixed-methods feasibility study protocol. BMJ Open. 2020 Nov 16;10(11):e041667. doi: 10.1136/bmjopen-2020-041667. PMID 33199427
- [Background] Gordon TC, Kemp AH, Edwards DJ. Mixed-methods feasibility outcomes for a novel ACT-based video game 'ACTing Minds' to support mental health. BMJ Open. 2024 Mar 29;14(3):e080972. doi: 10.1136/bmjopen-2023-080972. PMID 38553053